CLINICAL TRIAL: NCT06978933
Title: A Prospective, Exploratory Study to Evaluate the Safety and Efficacy of the Combination of ABSK-011 and ABSK043 in Patients With Previously Treated Unresectable or Metastatic Hepatocellular Carcinoma With FGF19 Overexpression
Brief Title: FGF19 Overexpression Combination Unified Study in HCC-19
Acronym: FOCUS-19
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSK-011-2002-IIT
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABSK-011+ABSK043 (Experimental)
  Interventions: Drug: ABSK-011

INTERVENTIONS:
Drug: ABSK-011 — Drug: ABSK-011 RP2D according to the results of Phase I trial
  Other Names:
  • FGFR4 inhibitor Drug: ABSK043 RP2D according to the results of Phase I trial
  Other Names:
  • Oral PD-L1 inhibitor

SUMMARY:
This study is designed prospectively to investigate the safety and efficacy of ABSK-011 and ABSK043 in patients with previously treated unresectable or metastatic hepatocellular carcinoma (HCC) harboring FGF19 overexpression. ABSK-011, an oral, selective FGFR4 inhibitor which can irreversibly bind to the target. ABSK043, is an orally available, selective and potent inhibitor targeting the interaction of PD-1 and PD-L1, Safety, tolerability, and preliminary efficacy of ABSK-011 or ABSK043 were explored in a phase 1 trial ABSK-011-101 (NCT04906434) and ABSK043-101 (NCT04964375) trial, respectively. This trial focuses on the efficacy of the combination of ABSK-011 and ABSK043 in patients with previously treated unresectable or metastatic HCC harboring FGF19 overexpression.

DETAILED DESCRIPTION:
The patients that meet the Inclusion and Exclusion Criteria will treat with ABSK-011 RP2D and ABSK043 RP2D until the disease progression

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HCC confirmed by pathological histology or cytology, or meeting the clinical diagnostic criteria for HCC as the AASLD or Guidelines for the diagnosis and treatment of primary liver cancer (China).
2. Progression of disease confirmed by imaging after receiving at least one line of systemic therapy
3. The central laboratory test report for FGF19 overexpression positive.
4. ECOG performance status of 0 or 1;
5. Adequate organ and marrow function defined by study-specified laboratory tests;

Exclusion Criteria:

1. Has received prior therapy with FGFR4 or pan-FGFR inhibitors;
2. Hypersensitivity for any constituent of ABSK-011 or ABSK043;
3. Past or current hepatic encephalopathy; patients with known untreated or inadequately controlled central nervous system metastases that have not been effectively managed with treatment
4. have other malignant tumors that are currently in a progressive stage or require effective treatment
5. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the objective response rate of ABSK-011 plus ABSK043 in patients with previously treated unresectable or metastatic HCC harboring FGF19 overexpression | 10 months
  Objective response rate (ORR): complete response and partial response determined by the investigator according to RECIST v1.1 and to be confirmed

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xia, MD, Study Chair — Shanghai Jiao Tong University school of medicine affiliate Renji Hospital; Hao Feng, Ph.D.,MD, Principal Investigator — Shanghai Jiao Tong University school of medicine affiliate Renji Hospital
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No